CLINICAL TRIAL: NCT01004770
Title: An Intravenous, Single Dose Safety, Tolerance and Pharmacokinetic Study of GE-145 in Healthy Volunteers Undergoing a Contrast-enhanced Abdominal Computed Tomography (CT) Scan
Brief Title: Single Dose Safety, Tolerance and Pharmacokinetic Study in Healthy Volunteers Undergoing Contrast-enhanced Abdominal Computed Tomography (CT)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: Medpace, Inc. (Industry); i3 Statprobe (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GE-145-001
Record Dates: First submitted 2009-10-23; First posted 2009-10-30 (Estimated); Results first posted 2012-04-04 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
Keywords: CECT - Contrast-enhanced computed tomography; HCG - Human Chorionic Gonadotropin; HU - Hounsfield Units; Patient Safety; Tolerance; Pharmacokinetic
MeSH Terms: interventions — 5-(formyl-(3-(formyl-(3,5-bis (2,3-dihydroxypropylcarbamoyl)-2,4,6-triiodophenyl) amino)-2-hydroxypropyl)amino)-N,N'-bis(2,3-dihydroxypropyl)-2,4,6-triiodobenzene-1,3-dicarboxamide; Injections; iodixanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (AH113111 Injection) (Experimental)
  Interventions: Drug: GE-145 (AN113111) Injection
- 2 (Visipaque Injection) (Active Comparator): An additional 10 subjects will receive Visipaque (iodixanol) 320 mg I/mL) at a dose of 450 mg/kg.
  Interventions: Drug: Visipaque (iodixanol) Injection

INTERVENTIONS:
Drug: GE-145 (AN113111) Injection — 40 healthy volunteers (10 per treatment group) will receive AH113111 320 mg I/mL at 1 of 4 possible doses (300, 450, 600, or 900 mg I/kg) as a single intravenous (IV) administration.
  Other Names: AH113111; GE-145
  Arms: 1 (AH113111 Injection)
Drug: Visipaque (iodixanol) Injection — An additional 10 subjects will receive Visipaque (iodixanol) 320 mg I/mL) at a dose of 450 mg/kg.
  Other Names: Visipaque; Iodixanol
  Arms: 2 (Visipaque Injection)

SUMMARY:
This is a non-randomized dose-escalating study that will evaluate the safety and tolerability of GE-145 at four different dose levels through the assessment of clinical laboratories, vital signs, physical examinations, electrocardiograms (ECGs) and the frequency and intensity of adverse events (AEs). It will characterize the pharmacokinetic properties of GE-145 through the evaluation of serum and urine. It will evaluate the radiographic density in regions of interest (ROI) and the overall diagnostic quality following administration of GE-145.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females between 18 and 60 years of age.
* For women who are either surgically sterile or are postmenopausal, enrollment in the study without a pregnancy test at screening will be allowed. For women of childbearing potential, the results of a serum and urine HCG pregnancy test (with the result known on the day of and before IMP administration) must be negative.
* Subjects are able and willing to comply with study procedures and sign an informed consent.

Exclusion Criteria:

* Known history of a reaction to any iodinated-based contrast agent or with multiple allergies (i.e. foods, pets, medications, etc).
* Subjects receiving any medication for which the use of an iodinated contrast agent is contraindicated (i.e.. metformin).
* Subjects with suspicion or diagnosis of hyperthyroidism.
* Women that are breastfeeding at the screening and/or enrolment period.
* Usage of any non-FDA-approved pharmaceutical or therapy within 30 days prior to screening or enrolment in another clinical study within 30 days prior to screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2009-10; Primary Completion 2010-02 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rubin Sheng, MD, Study Director — GE Healthcare
Locations (1):
- GE Healthcare, Princeton, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- GE-145 Injection-300mg of Iodine/mL: GE-145 x 300 milligram (mg) Iodine (I)/mL at doses of 300mgI/kg. The subjects in each dose group only received one dose.
- GE-145 Injection-450mg of Iodine/mL: GE-145 x 450 milligram (mg) Iodine (I)/mL a doses of 450mgI/kg. The subjects in each dose group only received one dose.
- GE-145 Injection-600mg of Iodine/mL: GE-145 x 600 milligram (mg) Iodine (I)/mL a doses of 600mgI/kg. The subjects in each dose group only received one dose.
- GE-145 Injection-900mg of Iodine/mL: GE-145 x 900 milligram (mg) Iodine (I)/mL a doses of 900mgI/kg. The subjects in each dose group only received one dose.
- Visipaque Injection: Visipaque x 320mgI/mL at a dose of 450mgI/kg
Period: Overall Study
Arm/Group | GE-145 Injection-300mg of Iodine/mL | GE-145 Injection-450mg of Iodine/mL | GE-145 Injection-600mg of Iodine/mL | GE-145 Injection-900mg of Iodine/mL | Visipaque Injection
Started | 10 | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GE-145 Injection-300mg of Iodine/mL | GE-145 Injection-450mg of Iodine/mL | GE-145 Injection-600mg of Iodine/mL | GE-145 Injection-900mg of Iodine/mL | Visipaque Injection | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 10 | 10 | 50
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 26.5 (3.89) | 27.2 (11.54) | 30.8 (11.50) | 27.4 (10.05) | 31.3 (11.91) | 28.6 (10.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 9 | 3 | 2 | 19
  Male | 8 | 7 | 1 | 7 | 8 | 31
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 10 | 10 | 50

OUTCOME MEASURES:

1. Primary Outcome: Blood Urea Nitrogen and Creatinine Serum Values
Description: Blood Urea Nitrogen and Creatinine serum value results taken up to and including 72 hours.
Time Frame: Baseline and up to and including 72 hours post contrast administration
Population: Per Study Protocol
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | GE-145 Injection-300mg of Iodine/mL | GE-145 Injection-450mg of Iodine/mL | GE-145 Injection-600mg of Iodine/mL | GE-145 Injection-900mg of Iodine/mL | Visipaque Injection
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
mg/dL
  Blood Urea Nitrogen (BUN) - Baseline | 12.3 (3.2) | 14.7 (3.0) | 14.5 (4.3) | 12.8 (4.5) | 11.9 (4.6)
  BUN - 8 h post | 10.8 (3.1) | 14.2 (2.8) | 14.7 (6.5) | 11.8 (4.7) | 12.4 (2.5)
  BUN - 24 h post | 11.1 (3.0) | 14.0 (2.9) | 12.5 (3.2) | 11.5 (3.3) | 11.2 (2.1)
  BUN - 48 h post | 11.7 (3.1) | 14.8 (2.4) | 13.7 (4.7) | 12.4 (3.8) | 11.3 (3.4)
  BUN - 72 h post | 12.2 (2.3) | 14.2 (2.8) | 14.9 (4.6) | 12.5 (3.7) | 12.5 (4.2)
  Creatinine - Baseline | 0.79 (0.19) | 0.79 (0.15) | 0.64 (0.10) | 0.87 (0.20) | 0.81 (0.15)
  Creatinine - 8 h post | 0.76 (0.19) | 0.82 (0.12) | 0.64 (0.11) | 0.83 (0.19) | 0.79 (0.14)
  Creatinine - 24 h post | 0.75 (0.19) | 0.78 (0.13) | 0.61 (0.10) | 0.76 (0.16) | 0.78 (0.16)
  Creatinine - 48 h post | 0.76 (0.21) | 0.78 (0.15) | 0.62 (0.11) | 0.88 (0.23) | 0.81 (0.17)
  Creatinine - 72 h post | 0.78 (0.15) | 0.74 (0.13) | 0.64 (0.13) | 0.82 (0.20) | 0.85 (0.14)

2. Primary Outcome: Vital Signs (Blood Pressure) Systolic and Diastolic Values
Description: Systolic and Diastolic bolld pressure taken up to and including 8 hours
Time Frame: Baseline and up to and including 8 hours post contrast administation.
Population: Per Study Protocol
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | GE-145 Injection-300mg of Iodine/mL | GE-145 Injection-450mg of Iodine/mL | GE-145 Injection-600mg of Iodine/mL | GE-145 Injection-900mg of Iodine/mL | Visipaque Injection
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
mm Hg
  Systolic BP - Baseline | 113.1 (10.87) | 125.5 (13.10) | 116.3 (11.49) | 114.9 (12.98) | 118.1 (12.15)
  Systolic BP - 10 min post | 110.6 (6.88) | 123.4 (8.32) | 115.3 (11.73) | 112.2 (13.31) | 118.0 (5.35)
  Systolic BP - 20 min post | 114.2 (8.51) | 121.8 (11.44) | 120.4 (5.78) | 112.6 (10.59) | 120.0 (4.99)
  Systolic BP - 1 h post | 110.4 (9.65) | 120.5 (7.59) | 115.7 (11.13) | 112.7 (10.14) | 115.6 (9.00)
  Systolic BP - 8 h post | 113.6 (11.19) | 116.6 (16.60) | 99.0 (8.76) | 110.1 (10.69) | 115.3 (13.94)
  Diastolic BP - Baseline | 71.7 (9.32) | 72.5 (12.33) | 74.3 (9.03) | 69.9 (12.48) | 77.2 (9.52)
  Diastolic BP - 10 min post | 69.4 (9.65) | 74.3 (8.25) | 73.3 (10.52) | 70.4 (11.05) | 76.0 (9.83)
  Diastolic BP - 20 min post | 69.6 (8.47) | 70.8 (10.17) | 75.0 (7.06) | 71.8 (10.26) | 77.1 (7.31)
  Diastolic BP - 1 h post | 67.4 (10.54) | 70.0 (5.79) | 70.4 (7.63) | 72.2 (7.50) | 72.2 (8.63)
  Diastolic BP - 8 h post | 70.4 (8.58) | 70.1 (10.96) | 64.5 (5.32) | 69.0 (5.60) | 68.8 (10.96)

3. Primary Outcome: Vital Sign (Heart Rate in Beats Per Minute-(Bpm)) Values
Description: Heart Rate (beats per minute-(bpm)) taken up to and including 8 hours.
Time Frame: Baseline and up to and including 8 hours post contrast administration
Population: Per Study Protocol
Measure: Mean (Standard Deviation); unit: > 10 beats per minute (bpm)
Arm/Group | GE-145 Injection-300mg of Iodine/mL | GE-145 Injection-450mg of Iodine/mL | GE-145 Injection-600mg of Iodine/mL | GE-145 Injection-900mg of Iodine/mL | Visipaque Injection
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
> 10 beats per minute (bpm)
  Heart Rate - Baseline | 65.8 (8.35) | 76.0 (11.53) | 77.9 (6.23) | 75.9 (15.00) | 86.1 (7.40)
  Heart Rate - 10 min post | 64.1 (9.78) | 75.7 (11.36) | 77.1 (10.38) | 78.6 (10.17) | 86.7 (8.74)
  Heart Rate - 20 min post | 65.0 (10.85) | 76.0 (12.41) | 75.4 (5.10) | 75.9 (9.70) | 87.4 (8.54)
  Heart Rate - 1 h post | 65.1 (8.67) | 73.9 (8.60) | 72.5 (9.89) | 77.3 (9.87) | 78.5 (10.84)
  Heart Rate - 8 h post | 69.1 (11.06) | 71.1 (15.89) | 75.2 (9.39) | 75.2 (12.04) | 79.4 (13.27)

4. Primary Outcome: 12-Lead Electrocardiogram (ECG) Values
Description: 12-Lead ECG values taken up to and including 24 hours
Time Frame: Baseline and up to and including 24 hours post contrast administration
Population: Per Study Protocol
Measure: Mean (Standard Deviation); unit: QTcB (msec)
Arm/Group | GE-145 Injection-300mg of Iodine/mL | GE-145 Injection-450mg of Iodine/mL | GE-145 Injection-600mg of Iodine/mL | GE-145 Injection-900mg of Iodine/mL | Visipaque Injection
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
QTcB (msec)
  ECG - Baseline | 408.6 (24.3) | 420.2 (21.2) | 425.0 (17.9) | 410.2 (20.8) | 435.6 (17.8)
  ECG - 20 min post | 413.5 (18.4) | 422.9 (22.1) | 434.0 (14.2) | 418.2 (22.9) | 418.7 (24.6)
  ECG - 24 h post | 412.6 (15.4) | 411.4 (21.7) | 430.5 (18.8) | 401.5 (22.2) | 424.4 (19.0)

5. Primary Outcome: Radiographic Density of the Region of Interest (ROI) Between Pre and Post Contrast Image
Description: Radiographic Density differences of the abdominal aorta, pre and post contrast on the Arterial Phase
Time Frame: Pre and post contrast administration
Population: Per Study Protocol
Measure: Mean (Standard Deviation); unit: Hounsfield Units
Arm/Group | GE-145 Injection-300mg of Iodine/mL | GE-145 Injection-450mg of Iodine/mL | GE-145 Injection-600mg of Iodine/mL | GE-145 Injection-900mg of Iodine/mL | Visipaque Injection
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Hounsfield Units
  Abdominal aorta-Pre-Contrast | 39.8 (5.87) | 44.0 (5.83) | 44.7 (4.21) | 43.9 (3.56) | 44.5 (7.01)
  Abdominal aorta-Post-Contrast | 243.8 (41.78) | 263.6 (78.60) | 301.6 (74.96) | 305.8 (52.64) | 245.8 (45.69)

ADVERSE EVENTS:
Time Frame: 7 Day Followup
Arm/Group | GE-145 Injection-300mg of Iodine/mL | GE-145 Injection-450mg of Iodine/mL | GE-145 Injection-600mg of Iodine/mL | GE-145 Injection-900mg of Iodine/mL | Visipaque Injection
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 2/10 | 1/10 | 0/10 | 0/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GE-145 Injection-300mg of Iodine/mL (N=10) | GE-145 Injection-450mg of Iodine/mL (N=10) | GE-145 Injection-600mg of Iodine/mL (N=10) | GE-145 Injection-900mg of Iodine/mL (N=10) | Visipaque Injection (N=10)
Radiation Exposure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Patient received radiation exposure
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GE-145 Injection-300mg of Iodine/mL (N=10) | GE-145 Injection-450mg of Iodine/mL (N=10) | GE-145 Injection-600mg of Iodine/mL (N=10) | GE-145 Injection-900mg of Iodine/mL (N=10) | Visipaque Injection (N=10)
Skin (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No